CLINICAL TRIAL: NCT04991454
Title: Xenon MRI in Pulmonary Hypertension
Brief Title: Xenon MRI Pulm Hypertension
Acronym: Jupiter PH
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Bastiaan Driehuys (Other)
Responsible Party: Sponsor-Investigator, Bastiaan Driehuys, Associate Professor of Radiology, Duke University
Organization: Duke University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00107613
Record Dates: First submitted 2021-07-07; First posted 2021-08-05 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-07

CONDITIONS: Pulmonary Hypertension; Pulmonary Arterial Hypertension
Keywords: Lung Transplant; Xenon; MRI
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Arterial Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- end-stage pulmonary hypertension . (Other): subjects with end-stage PH that currently on the waitlist for lung transplant
  Interventions: Drug: 129Xe Hyperpolarized
- following pulmonary arterial hypertension subjects (Other): Following pulmonary arterial hypertension subjects upto 24 months
  Interventions: Drug: 129Xe Hyperpolarized

INTERVENTIONS:
Drug: 129Xe Hyperpolarized — Each xenon dose will be limited to a volume less than 25% of subject lung capacity (TLC), as is the case for all protocols currently carried out under IND 109,490.

SUMMARY:
The overall objective outlined in this study is to determine how pulmonary vascular remodeling in PAH at a cellular and pathological level is associated with changes in gas exchange physiology and hemodynamics (monitored with 129Xe MRI/MRS) and how these signals change with disease progression or treatment.

DETAILED DESCRIPTION:
In aim 1, the study team will compare 129Xe MRI signatures to lung explant pathology, cellular identity from single-cell RNA sequencing, and cellular phenotypes in gas exchange defects to areas that are spared, which the team will hypothesize are exposed to lower levels of hemodynamic shear stress. This will be done by performing 129Xe MRI scans in fifteen subjects (cohort 1) with PAH awaiting a lung transplant, followed by a pathologic assessment (with usual histopathology and single cell RNA sequencing) of the subject's explanted lung after transplant. The study team expect that areas of proliferation and fibrosis will correlate with 129Xe MRI gas exchange and spectroscopic defects

In aim 3, The study team will test whether directly monitoring lung pathology with 129Xe MRI will provide additional prognostic information to standard-of-care clinical monitoring in 45 subjects (cohort 2). At 6-month follow-up appointments, standard-of-care assessments including labs, echocardiography, and six-minute walk distance and 129Xe MRI will be collected. The study team expect that In aim 1, the study team will compare 129Xe MRI signatures to lung explant pathology, cellular identity from single-cell RNA sequencing, and cellular phenotypes in gas exchange defects to areas that are spared, which the study team hypothesizes are exposed to lower levels of hemodynamic shear stress. This will be done by performing 129Xe MRI scans in fifteen subjects (cohort 1) with PAH awaiting a lung transplant, followed by a pathologic assessment (with usual histopathology and single-cell RNA sequencing) of the subject's explanted lung after transplant. The study team expect that areas of proliferation and fibrosis will correlate with 129Xe MRI gas exchange and spectroscopic defects

ELIGIBILITY:
Inclusion Criteria of Cohort 1

Subjects must meet all of the following inclusion criteria to be eligible for enrollment into the trial:

1. Outpatients of either gender, Age 18-75
2. Awaiting a lung transplant
3. Diagnosis of precapillary PH (right heart catheterization demonstrating hemodynamic criteria of a mean pulmonary artery pressure (mPAP) ≥ 25 mmHg, pulmonary vascular resistance ≥ 3 WU, pulmonary capillary wedge pressure ≤ 15 mmHg) in the setting of Group 1 (PAH), 3 (PH due to chronic lung disease, 4 (PH due to pulmonary artery obstructions), or 5 (PH due to miscellaneous causes)
4. Willing and giving informed consent and adhere to visit/protocol schedules (consent must be given before any study procedures are performed).
5. Women of childbearing potential must have a negative urine pregnancy test before MRI

Exclusion Criteria of Cohort 1

Subjects presenting with any of the following will not be included in the trials:

1. Moderate to severe heart disease (LVEF <45%, Severe LV hypertrophy, Moderate to severe valvular disease)
2. PH due to schistosomiasis
3. Active cancer
4. Sickle cell anemia
5. Prisoners and pregnant women will not be approached for the study
6. Conditions that will prohibit MRI scanning (metal in eye, claustrophobia, inability to lie supine)
7. Medical or psychological conditions which, in the opinion of the investigator, might create undue risk to the subject or interfere with the subject's ability to comply with the protocol requirements

Inclusion Criteria of Cohort 2

Subjects must meet all of the following inclusion criteria to be eligible for enrollment into the trial:

1. Treatment naïve or treatment started within the last 3 months
2. Outpatients of either gender, Age 18-75
3. WHO functional class (FC) 2-3 symptoms with a diagnosis of group 1 PH (mean pulmonary artery pressures (mPAP) > 20 mmHg, pulmonary capillary wedge pressure (PCWP) ≤ 15mmHg and pulmonary vascular resistance (PVR) ≥3 WU)
4. Willing and able to give informed consent and adhere to visit/protocol schedules (consent must be given before any study procedures are performed).
5. Women of childbearing potential must have a negative urine pregnancy test before MRI

Exclusion Criteria of Cohort 2

Subjects presenting with any of the following will not be included in the trials:

1. Sarcoidosis
2. Active cancer
3. Sickle cell anemia
4. Liver disease (Childs-Pugh class C)
5. Any conditions that prevent the performance of 129Xe MRI scans.
6. Prisoners and pregnant women will not be approached for the study.
7. Conditions that will prohibit MRI scanning (metal in eye, claustrophobia, inability to lie supine).
8. Medical or psychological conditions which, in the opinion of the investigator, might create undue risk to the subject or interfere with the subject's ability to comply with the protocol requirements

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
pulmonary vascular remodeling | 5 years
  The study team will determine whether the correlation between Red Blood Cell Signal from Xenon MRI to pathologic scoring of pulmonary vascular remodeling from histopathology is statistically significant.
Red Blood Cell Signal from Xenon MRI | 5 years
  We will determine whether the correlation between Red Blood Cell Signal from Xenon MRI to six minute walk distance, tricuspid annular plane excursion and right ventricular systolic pressure in longitudinal follow-up of PAH patients is statistically significant.

CONTACTS AND LOCATIONS:
Overall Officials: Sudarshan Rajagopal, MD, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No